CLINICAL TRIAL: NCT06730295
Title: Elimination of PTV Margins Based on Online Adaptive Stereotactic Radiotherapy for Centrally Located Early-stage Non-small Cell Lung Cancer: a Prospective, Single-arm, Phase II Study
Brief Title: Elimination of PTV Margins Based on Online Adaptive Stereotactic Radiotherapy for Centrally Located Early-stage Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Pro., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10122
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer (NSCLC)
Keywords: lung cancer; radiotherapy; early stage
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The study group (Experimental): Patients in the study group will receive online adaptive stereotactic body radiotherapy (without PTV expansion margin). The total dose will be 39-42Gy/3fractions, administered once daily. Both FBCT and 4DCT will be acquired before initiating treatment at each fraction.
  Interventions: Radiation: Online adaptive SBRT

INTERVENTIONS:
Radiation: Online adaptive SBRT — Online adaptive SBRT (without PTV expansion margin). The total dose will be 39-42Gy/3 fractions, administered once daily. FBCT and 4DCT will be acquired.

SUMMARY:
This study aims to explore the safety and efficacy of eliminating the PTV (planning target volume) margins based on online adaptive stereotactic radiotherapy for patients with centrally located early-stage non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed untreated early-stage non-small cell lung cancer (T1-2N0M0), or recurrent disease (rT1-2N0M0) that is inoperable or where the patient is unwilling to undergo surgery.
* Centrally located lung cancer.
* Age 18 years or older, regardless of gender.
* ECOG performance status score of 0-2.
* Serum hemoglobin ≥ 80 g/L, platelets ≥ 100,000/μL, absolute neutrophil count ≥ 1,500/μL.
* Serum creatinine ≤ 1.25 times the upper normal limit (UNL) or creatinine clearance ≥ 60 ml/min.
* Serum bilirubin ≤ 1.5 times UNL, AST (SGOT) and ALT (SGPT) ≤ 2.5 times UNL, alkaline phosphatase ≤ 5 times UNL.
* FEV1 ≥ 0.5 L.
* Normal CB6 range.
* The patient and their family agree and sign the informed consent form.

Exclusion Criteria:

* Any other disease or condition that contraindicates radiotherapy (e.g., active infections, within 6 months post-myocardial infarction, symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmias).
* Pregnant or breastfeeding women, women who have not undergone pregnancy testing, and pregnant individuals.
* Individuals with substance abuse issues, chronic alcoholism, or AIDS.
* Individuals with uncontrollable seizures or loss of self-control due to psychiatric disorders.
* Individuals with a history of severe allergies or specific sensitivities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher SBRT-related toxicity | 1-year
  Incidence of grade 3 or higher SBRT-related toxicity

SECONDARY OUTCOMES:
Objective response rate | 2 months after radiotherapy]
  Objective Response Rate (ORR) is defined as the proportion of patients whose tumor size decreases to a pre-specified value and is maintained for a certain period of time during cancer treatment. It includes the number of patients with Complete Response (CR) and Partial Response (PR) as a percentage of the total number of evaluable cases.
Local control rate | 2-year
  The control of the local lesion after treatment.
Progression-free survival | 2-year
  PFS measures the time from the start date of SBRT to disease progression, death from any cause or last follow up if alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haasbeek CJ, Lagerwaard FJ, Slotman BJ, Senan S. Outcomes of stereotactic ablative radiotherapy for centrally located early-stage lung cancer. J Thorac Oncol. 2011 Dec;6(12):2036-43. doi: 10.1097/JTO.0b013e31822e71d8. PMID 21892102
- [Background] Meng Y, Luo W, Xu H, Wang W, Zhou S, Tang X, Li Z, Zhou C, Yang H. Adaptive intensity-modulated radiotherapy with simultaneous integrated boost for stage III non-small cell lung cancer: Is a routine adaptation beneficial? Radiother Oncol. 2021 May;158:118-124. doi: 10.1016/j.radonc.2021.02.019. Epub 2021 Feb 23. PMID 33636232
- [Background] Verma V, Shostrom VK, Kumar SS, Zhen W, Hallemeier CL, Braunstein SE, Holland J, Harkenrider MM, S Iskhanian A, Neboori HJ, Jabbour SK, Attia A, Lee P, Alite F, Walker JM, Stahl JM, Wang K, Bingham BS, Hadzitheodorou C, Decker RH, McGarry RC, Simone CB 2nd. Multi-institutional experience of stereotactic body radiotherapy for large (>/=5 centimeters) non-small cell lung tumors. Cancer. 2017 Feb 15;123(4):688-696. doi: 10.1002/cncr.30375. Epub 2016 Oct 14. PMID 27741355
- [Background] Bezjak A, Paulus R, Gaspar LE, Timmerman RD, Straube WL, Ryan WF, Garces YI, Pu AT, Singh AK, Videtic GM, McGarry RC, Iyengar P, Pantarotto JR, Urbanic JJ, Sun AY, Daly ME, Grills IS, Sperduto P, Normolle DP, Bradley JD, Choy H. Safety and Efficacy of a Five-Fraction Stereotactic Body Radiotherapy Schedule for Centrally Located Non-Small-Cell Lung Cancer: NRG Oncology/RTOG 0813 Trial. J Clin Oncol. 2019 May 20;37(15):1316-1325. doi: 10.1200/JCO.18.00622. Epub 2019 Apr 3. PMID 30943123
- [Background] Adebahr S, Collette S, Shash E, Lambrecht M, Le Pechoux C, Faivre-Finn C, De Ruysscher D, Peulen H, Belderbos J, Dziadziuszko R, Fink C, Guckenberger M, Hurkmans C, Nestle U. LungTech, an EORTC Phase II trial of stereotactic body radiotherapy for centrally located lung tumours: a clinical perspective. Br J Radiol. 2015 Jul;88(1051):20150036. doi: 10.1259/bjr.20150036. Epub 2015 Apr 15. PMID 25873481
- [Background] Sun B, Brooks ED, Komaki RU, Liao Z, Jeter MD, McAleer MF, Allen PK, Balter PA, Welsh JD, O'Reilly MS, Gomez D, Hahn SM, Roth JA, Mehran RJ, Heymach JV, Chang JY. 7-year follow-up after stereotactic ablative radiotherapy for patients with stage I non-small cell lung cancer: Results of a phase 2 clinical trial. Cancer. 2017 Aug 15;123(16):3031-3039. doi: 10.1002/cncr.30693. Epub 2017 Mar 27. PMID 28346656
- [Background] Prezzano KM, Ma SJ, Hermann GM, Rivers CI, Gomez-Suescun JA, Singh AK. Stereotactic body radiation therapy for non-small cell lung cancer: A review. World J Clin Oncol. 2019 Jan 10;10(1):14-27. doi: 10.5306/wjco.v10.i1.14. PMID 30627522